CLINICAL TRIAL: NCT06464887
Title: Construction and Validation of an Early Prediction Nomogram for Recurrent Acute Pancreatitis Based on the MIMIC Database
Brief Title: A Predictive Model for Recurrent Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Qinghao Wang (Other)
Responsible Party: Sponsor-Investigator, Qinghao Wang, Master of Medicine, Yangzhou University
Organization: Yangzhou University (Other)
Other Study IDs: 20200047
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Acute Pancreatitis
Keywords: Recurrent acute pancreatitis; Prediction
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent acute pancreatitis
- Non-recurrent acute pancreatitis

SUMMARY:
The goal of this observational study is to learn about recurrent acute pancreatitis (RAP) .The main questions it aims to answer are:

1. What are the risk factors for RAP?
2. How to predict RAP?

All patients with acute pancreatitis will be given standardized treatment for the condition.

The researchers will compare the RAP group with the non-RAP group to find the risk factors for RAP.

DETAILED DESCRIPTION:
Investigators retrospectively collected data from the Medical Information Mart for Intensive Care-IV (MIMIC-IV) database and from patients with acute pancreatitis (AP) in the Department of Gastroenterology of Clinical Medical College of Yangzhou University between January 2016 and December 2017, forming the primary and validation cohort, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of acute pancreatitis (AP)
* Age ≥18 years
* Systematic examination and diagnostic information were available after admission

Exclusion Criteria:

* Not the first episode of AP
* The duration of hospital stay was less than 24 hours
* Died within the first episode of AP
* A history of chronic pancreatitis or tumor
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We collected data from the Medical Information Mart for Intensive Care-IV (MIMIC-IV) database and from patients with acute pancreatitis in the Department of Gastroenterology of Clinical Medical College of Yangzhou University between January 2016 and December 2017, forming the primary and validation cohort, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 659 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience Recurrent Acute Pancreatitis | From admission to 3 years after discharge.
  Recurrent acute pancreatitis was defined as two or more confirmed episodes of acute pancreatitis, excluding chronic pancreatitis, with an interval of more than 3 months between attacks, and complete resolution of symptoms during the inter-episodic periods.

REFERENCES:
- [Background] Johnson AEW, Bulgarelli L, Shen L, Gayles A, Shammout A, Horng S, Pollard TJ, Hao S, Moody B, Gow B, Lehman LH, Celi LA, Mark RG. MIMIC-IV, a freely accessible electronic health record dataset. Sci Data. 2023 Jan 3;10(1):1. doi: 10.1038/s41597-022-01899-x. PMID 36596836
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216